CLINICAL TRIAL: NCT01455740
Title: A Commitment Device for Medication Adherence Among HIV Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0005
Record Dates: First submitted 2011-10-13; First posted 2011-10-20 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV
Keywords: Acquired Immunodeficiency Syndrome; HIV; Commitment; Financial Incentives
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The study used a randomized trial design for two treatment arms: (i) Participants in the provider visit incentive (PVI) arm were told that they would receive $30 after attending each scheduled provider visit (a CCT). (ii) Participants in the incentive choice (IC) were given a choice between the above CCT and a commitment contract, which made the $30 payment conditional on the patient attending the provider visit and meeting an ART adherence threshold. A block randomization scheme, stratified on whether or no the majority of the participant's three previous viral load measurements were suppressed, assigned 21 individuals to the PVI arm and 19 to the IC arm.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Provider Visit Incentive (PVI) (Experimental): Participants were told that they would receive $30 after attending each scheduled provider visit (a CCT).
  A block randomization scheme, stratified on whether or not the majority of the participant's three previous viral load measurements were suppressed, assigned 21 individuals to the PVI arm.
  Interventions: Behavioral: Provider Visit Incentive (PVI)
- Incentive Choice (IC) (Experimental): Participants were given a choice between the CCT described in the PVI arm and a commitment contract, which made the $30 payment conditional on the patient attending the provider visit AND meeting an ART adherence threshold.
  A block randomization scheme, stratified on whether or not the majority of the participant's three previous viral load measurements were suppressed, assigned 19 individuals to the IC arm.
  Interventions: Behavioral: Incentive Choice (IC)
- Passive Control (PC) (No Intervention): The study also included 70 individuals in a PC arm, who did not receive financial incentives. Individuals in the PC arm were not enrolled in the randomized trial but met basic study eligibility criteria during the same time period.

INTERVENTIONS:
Behavioral: Provider Visit Incentive (PVI) — All participants received the standard of care (SOC), which included not only medical care but also a wide range of social services. In addition, participants in the PVI arm received financial incentives designed to motivate health-improving behaviors. After the initial study enrollment visit, participants in the PVI arm received a $30 payment each time they showed up as scheduled for one of their next four HIV primary care visits.
  Participants in the PVI arm were also asked to return for a sixth, unanticipated study visit approximately three months after the last of the four study visits to which the incentive scheme applied. To reduce attrition, participants were offered $100 for showing up to the fifth and sixth study visits.
  Arms: Provider Visit Incentive (PVI)
Behavioral: Incentive Choice (IC) — All participants received the SOC. In addition, participants in the IC arm received financial incentives designed to motivate health-improving behaviors. At the initial study enrollment visit, participants in the IC arm chose between either the incentive scheme assigned to the PVI arm or an incentive scheme that tied payments to clinic attendance and ART medication adherence. Participants who selected the 2nd option received a $30 payment at each of their next 4 HIV primary care visits if the (i) showed up as scheduled and (ii) presented a dose-recording pill bottle cap indicating that they correctly took at least 90% of doses of a sentinal medication since the previous study visit.
  Participants in the IC arm were also asked to return for a 6th, unanticipated study visit approximately three months after the last of the 4 study visits to which the incentive scheme applied. To reduce attrition, participants were offered $100 for showing up to the 5th and 6th study visits.
  Arms: Incentive Choice (IC)

SUMMARY:
We used a randomized trial design combined with a comparison to a non-randomized control group to study patients on appropriate antiretroviral therapy (ART) having virologic failure within a publicly-funded HIV clinic serving Atlanta, GA.

DETAILED DESCRIPTION:
This study demonstrated the feasibility of using commitment contracts in HIV care. Many previous interventions have produced statistically significant effects on ART adherence that do not persist after the intervention ends. A notable feature of our study is that after the incentives for ART adherence and provider visits were removed, participants who had been offered a commitment contract for ART adherence were more likely to achieve virologic suppression relative to individuals who had been assigned a conditional cash transfer for provider visits and relative to individuals who had been assigned the standard of care, although the difference was only statistically significant in the latter comparison. There were differences in the prevalence of missing outcomes across groups, but these differences were not statistically significant for the unanticipated post-incentive visit and therefore were unlikely to be the explanation for the results. Thus, financial rewards coupled with individual choice can increase engagement in healthy behaviors after incentives are removed.

ELIGIBILITY:
Inclusion Criteria:

* Attended the Grady Health System Infectious Disease Program (IDP)
* Most recent HIV-1 plasma RNA viral load (pVL) > 200 copies/mL; this value must have been measured within the prior 18 months and at least 6 months after starting the current ART regimen
* English-speaking

Exclusion Criteria:

* Using pillboxes
* Were planning to relocate
* Were enrolled in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Virologic Suppression (pVL =< 200 copies/mL) at Fifth Study Visit | 12 months (median)

SECONDARY OUTCOMES:
Virologic Suppression (pVL =< 200 copies/mL) at Unanticipated Sixth Study Visit | 15 months (median)

CONTACTS AND LOCATIONS:
Overall Officials: David I Laibson, Ph.D., Principal Investigator — National Bureau of Economic Research, Harvard University; Vincent Marconi, M.D., Principal Investigator — Emory University
Locations (1):
- Emory University Ponce Clinic, Atlanta, Georgia, United States

REFERENCES:
- [Result] Alsan M, Beshears J, Armstrong WS, Choi JJ, Madrian BC, Nguyen MLT, Del Rio C, Laibson D, Marconi VC. A commitment contract to achieve virologic suppression in poorly adherent patients with HIV/AIDS. AIDS. 2017 Jul 31;31(12):1765-1769. doi: 10.1097/QAD.0000000000001543. PMID 28514277